CLINICAL TRIAL: NCT07214701
Title: Sedative and Analgesic Effects of Dexmedetomidine Versus Ketamine in Patients Undergoing Varicocelectomy Under Spinal Anaesthesia: A Prospective Randomized Comparative Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed khalifa Mahmoud Saleh, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexmedet VS ketamine
Record Dates: First submitted 2025-10-05; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Varicocelectomy
MeSH Terms: interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): patiets received Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Group B (Active Comparator): patients receive Ketamine
  Interventions: Drug: Ketamine (0.5 mg/kg)

INTERVENTIONS:
Drug: Ketamine (0.5 mg/kg) — Intravenous infusion of ketamine 0.5 mg/kg over 10 minutes before spinal injection, diluted in 50 ml 0.9% NaCl Saline
  Arms: Group B
Drug: Dexmedetomidine — Intravenous infusion of dexmedetomidine 0.25 μg/kg over 10 minutes before spinal injection, diluted in 50 ml 0.9% NaCl Saline
  Arms: Group A

SUMMARY:
The demand for safe and effective sedation during spinal anesthesia has increased in recent years, particularly in ambulatory and minor surgical procedures. The ideal sedative agent should provide adequate anxiolysis and comfort, maintain cardiorespiratory stability, and allow rapid recovery without significant adverse effects .

Ketamine, a phencyclidine derivative, produces sedation, analgesia, and amnesia while maintaining airway reflexes and spontaneous respiration. However, it is often associated with undesirable psychomimetic reactions and sympathetic stimulation, including tachycardia and hypertension .

In contrast, dexmedetomidine, a highly selective α2-adrenergic agonist, provides cooperative sedation, analgesia, and reduced anesthetic requirements, but it may cause bradycardia and hypotension, particularly at higher doses .

The combination of ketamine and dexmedetomidine (often referred to as "Ketadex") has recently gained attention due to its synergistic effects. Evidence suggests that this combination improves hemodynamic stability, decreases emergence agitation, and provides superior analgesia compared to either agent alone [4,5]. Moreover, ketamine counteracts the bradycardia and hypotension induced by dexmedetomidine, while dexmedetomidine mitigates ketamine-induced psychomimetic side effects .

Despite these advantages, the optimal dosing regimen and comparative efficacy of the two drugs when used individually remain subjects of clinical debate. Recent randomized controlled trials comparing intravenous dexmedetomidine and ketamine during spinal anesthesia reported differences in sedation quality, hemodynamic stability, and recovery profile . Therefore, this study aims to compare the sedative and hemodynamic effects of intravenous dexmedetomidine versus ketamine infusion in patients undergoing varicocelectomy under spinal anesthesia.

the study aim to Compare sedative, analgesic efficacy, and safety profile of intravenous dexmedetomidine versus ketamine in patients undergoing varicocelectomy under spinal anaesthesia

ELIGIBILITY:
Inclusion Criteria:

* Age: from 18 to 40 years
* Sex: Male patients
* Operation: varicocelectomy under spinal anesthesia
* ASA physical states I-II

Exclusion Criteria:

* Psychiatric or neurological disorders
* Respiratory disorders
* Cardiovascular disorders
* Coagulation disorders
* Contraindications to neuraxial block (allergy to L.A, peripheral issues)
* spine deformity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
the time required in minutes to achieve OAA/S score 4. | 24 hour
  Modified observer's assessment of alertness/sedation score (OAA/S):
  5 Responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly and/or repeatedly 2 Responds only after mild prodding or shaking
  1 Responds only after painful stimulus 0 No response even after painful stimulus